CLINICAL TRIAL: NCT01611714
Title: Equity in Diagnostic Imaging Trial (EDIT)
Brief Title: Equity in Diagnostic Imaging Trial
Acronym: EDIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: GCO 02-0515(3); 3P60MD000270-09S1 (NIH)
Record Dates: First submitted 2012-04-13; First posted 2012-06-05 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Headache
Keywords: Racial/ethnic disparities; Imaging; Emergency; Headache
MeSH Terms: conditions — Headache; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Audit-feedback (Experimental): Arm 1: Audit-feedback only
  Interventions: Other: Audit-feedback
- CDS message (Experimental): Arm 2: CDS message only
  Interventions: Other: Clinical Decision Support
- Both Interventions (Experimental): Arm 3: Audit-feedback and CDS message
  Interventions: Other: Audit-feedback; Other: Clinical Decision Support
- Control (No Intervention): Arm 4: Control

INTERVENTIONS:
Other: Audit-feedback — Clinicians will receive a short email educational message at regular intervals alerting them to the historic disparities in diagnostic workup for SAH in our department and reminding them of the increased risk of SAH among African-American patients.
  Arms: Audit-feedback; Both Interventions
Other: Clinical Decision Support — Clinicians receive an embedded real-time Best Practice Alert (BPA) of increased rates of SAH among African-Americans when they open the "headache" electronic charting template.
  Other Names: CDS
  Arms: Both Interventions; CDS message

SUMMARY:
This study will 1) Develop two interventions: a) an audit-feedback email intervention that provides clinicians with data on CT scan ordering practices by patient race; and b) a clinical decision support (CDS) message in the electronic medical record headache template; and 2) Compare the effectiveness of these 2 interventions in eliminating a previously observed Black-White disparity in CT scanning rates to rule out subarachnoid hemorrhage (SAH).

DETAILED DESCRIPTION:
Investigators at our institution (Hwang & Richardson)* documented a racial disparity in the use of CT scans to diagnose subarachnoid hemorrhage, (SAH) a life-threatening form of stroke. Subsequent analyses found a similar finding in NHAMCS, a national ED Visit database*. The investigators will compare the effectiveness of 1) an audit-feedback intervention that provides data on race-specific CT rates and 2) a clinical decision support (CDS) message in the electronic "headache" charting template in eliminating the previously observed Black-White disparity in CT rates to rule out SAH.

Study Setting: The adult section of the Mount Sinai Emergency Department, an urban academic department with an annual volume of over 70,000 adult visits and a patient population representing a diverse cross-section of race and socioeconomic groups. The adult patients are cared for by a staff that includes: attending physicians, physician assistants, emergency medicine resident physicians, and rotating resident physicians from other specialties. The department has a dedicated CT scanner that is readily available around the clock. Epic Production is used for all physician and nurse documentation and for all order entry (including CT scans).

Over a 24-month period the investigators will compare the intervention and control groups' rates of testing for SAH across races, controlling for patient acuity, age and co-morbidities. Because the close working relationships among the attending and resident physicians in our department may lead to knowledge diffusion, the intervention may change the behavior of the control group as well as the intervention group, thus leading to an underestimation of the intervention effect as measured by the between- groups difference. The investigators will use a time series design to allow us to evaluate this effect. 10 months after the implementation of the first intervention, the clinical decision support message will be implemented. The impact of each intervention will be evaluated using a repeated measures design using a mixed linear model.

ELIGIBILITY:
Inclusion Criteria:

Attending Physicians, Emergency Room Resident Physicians, and PA's will be included if:

* they provide care to adult patients in the emergency department of Mount Sinai Hospital.

Patients will be enrolled for medical record review if

* they present with a complaint of headache and charted on the headache template in the period between four years pre-intervention and the end of the study period.

Exclusion Criteria:

* anyone who does not meet the inclusion criteria will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2010-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in CT usage rate | up to 24 months
  What is the impact of the email intervention, CDS intervention, and combined intervention on black-white difference in CT rates? A successful intervention should lead to a significant main effect for each experimental arm.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne D Richardson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States